CLINICAL TRIAL: NCT05744401
Title: A Multicenter, Long-term Extension Study to Evaluate the Safety, Tolerability, and Efficacy of AL002 in Participants With Alzheimer's Disease
Brief Title: A Long-term Extension Study to Evaluate Safety, Tolerability, and Efficacy of AL002 in Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Parent study failed to meet the primary endpoint and there were no treatment effects that favored AL002 on secondary clinical and functional endpoints.
Sponsor: Alector Inc. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL002-LTE
Record Dates: First submitted 2023-01-19; First posted 2023-02-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AL002 Dose 1 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002
- AL002 Dose 2 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002
- AL002 Dose 3 (Experimental): AL002 every 4 weeks
  Interventions: Drug: AL002

INTERVENTIONS:
Drug: AL002 — Administered via intravenous (IV) infusion

SUMMARY:
A long-term extension study to evaluate the safety, tolerability, and efficacy of AL002 in participants with Early Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a Phase 2, parallel-group, long-term extension (LTE), dose-blind study to evaluate the long-term safety and efficacy of AL002 in participants with Early Alzheimer's Disease. The study is a multicenter, global trial that will enroll participants who completed the planned treatment period in AL002-2 (parent study).

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Planned Treatment Period in the AL002-2 study.
* The participant is willing and able to give informed consent.
* Study partner who consents to study participation and who cares for/visits the participant at least 10 hours a week

Exclusion Criteria:

* Participants deemed not able to provide consent or assent by the Investigator or by local regulations.
* Participants who were prematurely and permanently discontinued from treatment in the parent study for safety reasons.
* Participation deemed inappropriate per Investigator discretion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by number of/incidence of Adverse Events (AEs), including AESI and SAEs. | Through study completion, up to 49 weeks
Safety and tolerability as measured by the number of incidence/MRI abnormalities. | Through study completion, up to 49 weeks

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, Principal Investigator
Locations (54):
- United States (15):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Charter Research, Lady Lake, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - Progressive Medical Research - ClinEdge - PPDS, Port Orange, Florida
  - Axiom Brain Health LLC, Tampa, Florida
  - "Alzheimers Research and Treatment Center-Wellington ", Wellington, Florida
  - Conquest Research LLC - Winter Park - ClinEdge - PPDS, Winter Park, Florida
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Advanced Clinical Institute, Neptune City, New Jersey
  - Feinstein Institute For Medical Research, Manhasset, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Summit Research Network, Portland, Oregon
- Argentina (2):
  - Instituto Privado Kremer, Córdoba, Córdoba Province
  - Centro de Psiquiatria Biologica, Mendoza
- Australia (3):
  - KaRa Institute of Neurological Disease, Macquarie Park, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Alfred Health, Melbourne, Victoria
- Canada (2):
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
- Germany (4):
  - Universitätsklinikum Ulm-Oberer Eselsberg 45, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, Munich, Bavaria
  - Ambulantes Gesundheitszebtrum der Charite GmbH, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
- Italy (10):
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome, Lazio
  - Azienda Policlinico Umberto, Rome, Lazio
  - Ospedale Isola Tiberina - Gemelli Isola, Rome, Lazio
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia, Lombardy
  - IRCCS - Centro S. Giovanni di Dio Fatebene fratelli, Brescia, Lombardy
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta-VIA MANGIAGALLI 3, Milan, Lombardy
  - ASL Biella - Ospedale degli Infermi, Ponderano, Piedmont
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico di Modena, Modena
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Brain Research Center Den Bosch - PPDS, 's-Hertogenbosch, North Brabant, Netherlands
- Poland (3):
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne NeuroProtect, Warsaw, Masovian Voivodeship
  - EUROMEDIS Sp. z o.o., Szczecin, West Pomeranian Voivodeship
- Spain (8):
  - Fundacion CITA Alzheimer Fundazioa, San Sebastián, Guipúzcoa
  - Centro De Atencion Especializada Oroitu, Getxo, Vizcaya
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Fundacion ACE Instituto Catalan de Neurociencias-Gran via de Carles III, 85 bis, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (6):
  - RE: Cognition Health - Plymouth, Plymouth, Devon
  - Re:Cognition Health - Guildford - PPDS, Guildford, Surrey
  - Re-Cognition Health - Bristol, Bristol
  - Re:Cognition Health, London
  - The National Hospital for Neurology and Neurosurgery, London
  - NeuroClin Glasgow, Motherwell